CLINICAL TRIAL: NCT05054933
Title: Feasibility and Safety of Ultrasound Capsule Endoscopy for Esophagus Examination：a Pilot Study
Brief Title: Ultrasound Capsule Endoscopy for Esophagus Examination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Professor, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Ultrasound CE
Record Dates: First submitted 2021-09-19; First posted 2021-09-23 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Esophageal Diseases
Keywords: capsule endoscopy; ultrasound
MeSH Terms: conditions — Esophageal Diseases | interventions — High-Energy Shock Waves; Endoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ultrasound capsule endoscopy examination (Other): Healthy volunteers or patients with suspected esophageal disease will be enrolled to take ultrasound capsule endoscopy examination followed by conventional endoscopic ultrasound examination within 2 weeks.
  Interventions: Other: ultrasound capsule endoscopy

INTERVENTIONS:
Other: ultrasound capsule endoscopy — Healthy volunteers or patients with suspected esophageal disease will be enrolled to take ultrasound capsule endoscopy examination followed by conventional endoscopic ultrasound examination within 2 weeks.

SUMMARY:
The aim of this pilot study is to assess the feasibility and safety of the clinical application of ultrasound capsule endoscopy in esophageal examination compared with conventional endoscopic ultrasound examination.

DETAILED DESCRIPTION:
Wireless capsule endoscopy has opened a new era by enabling remote diagnostic assessment of the gastrointestinal tract in a painless procedure. However, most commercially available devices only utilise optical imaging to examine the GI wall surface. Using this sensing modality, pathology within the GI wall cannot be detected. Micro-ultrasound (mUS) using high-frequency (>20 MHz) ultrasound can provide a means of transmural or cross-sectional image of the GI tract. Depth of imaging is approximately 10 mm with a resolution of between 40-120 μm that is sufficient to differentiate between subsurface histologic layers of the various regions of the GI tract. Ultrasound capsule endoscopy (USCE) uses a capsule equipped with mUS transducers that are capable of imaging below the GI wall surface, offering thereby a complementary sensing technique to optical imaging capsule endoscopy. In this work, a USCE device integrated with a 40 MHz ultrasonic transducer was developed to capture a full 360˚ image of the lumen. Previous animal studies of two anaesthetised Landrace pigs have demonstrated the effectiveness of the device. The reconstructed images demonstrate clear layer differentiation of the lumen wall. The tissue thicknesses measured from the B-scan images show good agreement with ex vivo images from the literature. The aim of this pilot study is to assess the feasibility and safety of the clinical application of ultrasound capsule endoscopy in esophageal examination compared with conventional endoscopic ultrasound examination.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 years or older.
2. Both inpatients and outpatients.
3. Healthy volunteers or patients with suspected esophageal disease
4. Able to provide informed consent.

Exclusion Criteria:

1. known or suspected complex history of gastrointestinal obstruction, stenosis or fistula.
2. dysphagia.
3. known or suspected possibility of active bleeding of digestive tract.
4. Pregnancy or suspected pregnancy..
5. Patients who have participated in or are participating in other clinical trials within three months.
6. Life-threatening conditions.
7. other circumstances that doctors consider inappropriate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-26 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of esophageal examination | 1 month
  Assess the success rate of the clinical application of ultrasound capsule endoscopy in esophageal examination, including observe the mucosa completely and obtain ultrasound cross-sectional images in specific parts.

SECONDARY OUTCOMES:
Diagnostic accuracy | 1 month
  The diagnostic accordance rate, sensitivity and specificity of lesions detected by ultrasound capsule endoscopy compared with conventional endoscopic ultrasound examination.
Clear layer differentiation of the esophageal wall structure | 1 month
  Assess the success rate of clear layer differentiation of the esophageal wall structure by ultrasound capsule endoscopy examination
Safety of ultrasound capsule endoscopy examination | 1 month
  The presence of any adverse events during ultrasound capsule endoscopy examination procedure will be recorded.
Examination time of esophagus | 1 month
  Record the time taken to finish examination of esophagus under ultrasound capsule endoscopy.
Discomfort scores associated with ultrasound capsule endoscopy examination | 1 month
  Assess the discomfort score caused by the string, swallowing the ultrasound capsule, pulling the capsule up or down, and pulling the capsule out. A visual analogue scale ranging from 0 (easy with no nausea) to 10 (very difficult or with sever nausea) was used to evaluate the degree of difficulty of the discomfort score caused by the string.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Professor, Principal Investigator — Changhai Hospital,Shanghai,China
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thosani N, Singh H, Kapadia A, Ochi N, Lee JH, Ajani J, Swisher SG, Hofstetter WL, Guha S, Bhutani MS. Diagnostic accuracy of EUS in differentiating mucosal versus submucosal invasion of superficial esophageal cancers: a systematic review and meta-analysis. Gastrointest Endosc. 2012 Feb;75(2):242-53. doi: 10.1016/j.gie.2011.09.016. Epub 2011 Nov 23. PMID 22115605
- [Background] Qiu Y, Huang Y, Zhang Z, Cox BF, Liu R, Hong J, Mu P, Lay HS, Cummins G, Desmulliez MPY, Clutton E, Zheng H, Qiu W, Cochran S. Ultrasound Capsule Endoscopy With a Mechanically Scanning Micro-ultrasound: A Porcine Study. Ultrasound Med Biol. 2020 Mar;46(3):796-804. doi: 10.1016/j.ultrasmedbio.2019.12.003. Epub 2020 Jan 3. PMID 31902446
- [Background] Ughi GJ, Gora MJ, Swager AF, Soomro A, Grant C, Tiernan A, Rosenberg M, Sauk JS, Nishioka NS, Tearney GJ. Automated segmentation and characterization of esophageal wall in vivo by tethered capsule optical coherence tomography endomicroscopy. Biomed Opt Express. 2016 Jan 8;7(2):409-19. doi: 10.1364/BOE.7.000409. eCollection 2016 Feb 1. PMID 26977350
- [Derived] Qiu XO, Jiang X, Chen YZ, Xia JS, Pan J, Wang L, Liao Z, Li ZS. New US capsule endoscopy for superficial and submucosal imaging of the esophagus: the first-in-human study. Gastrointest Endosc. 2023 Oct;98(4):642-652. doi: 10.1016/j.gie.2023.06.015. Epub 2023 Jun 24. PMID 37356634